CLINICAL TRIAL: NCT01342003
Title: HCV Genotype 1a Shows a Better Virological Response to Antiviral Therapy Than HCV Genotype 1b
Acronym: genotype
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera San Camillo Forlanini (Other)
Responsible Party: Adriano M Pellicelli, AO San Camillo Forlanini
Other Study IDs: 01
Record Dates: First submitted 2011-04-25; First posted 2011-04-26 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2010-10

CONDITIONS: Chronic Hepatitis C
Keywords: HCV infection; genotype 1a; genotype 1 b
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — HCVRNA determination was performed quantitatively before the treatment (TaqMan Roche Diagnostics). The TaqMan value utilized to determine the response was 15 IU/ml. TaqMan method was a standardized method utilized from December 2007 in all the center of the CLEO group. HCVRNA value was expressed as log10 IU/ml.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subtype 1a: subtype 1a patients treated with peginterferon plus ribavirin
- subtype 1b: subtype 1b patients treated with peginterferon plus ribavirin

SUMMARY:
Sustained virological response (SVR) to antiviral therapy in patients with chronic hepatitis C genotype 1 according to subtype (1a vs.1b) has not been extensively investigated. This observational study was carried out on a large group of "naïve" HCV patients to evaluate difference, if any, between HCV genotype 1 subtype 1a and 1b on the response to treatment with peginterferon (Peg-IFN) plus ribavirin.

DETAILED DESCRIPTION:
Despite the challenging perspective of the new antiviral drugs directly acting on hepatitis C viral replication such as protease and polymerase inhibitors, nowadays the standard treatment in genotype 1-chronic hepatitis C (CHC) is the combination of peghylated interferon (PEG-IFN) and ribavirin for 48 weeks. It has been extensively shown that patients infected with HCV genotype 1 have a lower rate of viral response than those infected with genotype 2 and 3. In large randomized multinational trials, sustained virological response (SVR) of around 50% has been obtained with peginterferon α2a plus ribavirin in the more difficult to treat subgroup of patients infected with HCV genotype 1. Furthermore, advanced fibrosis is a predictive factor of non response to antiviral treatment in genotype 1 virus [5-7]. Very few studies have evaluated SVR difference, if any, between subtypes 1a and 1b.

We have carried out an observational study on a large cohort of HCV "naïve" patients to evaluate the influence of HCV subtypes 1 on the response to treatment with Peg-INF plus ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* eligible subjects were naïve infected with HCV genotype 1 virus meeting the internationally recognised criteria for treatment (elevation of aminotransferases, inflammation and or fibrosis at liver biopsy).

Exclusion Criteria:

* infection with human immunodeficiency virus (HIV) or hepatitis B virus (HBV)
* alcohol intake greater than 20 gr daily
* the presence of active drug abuse, chronic systemic disease, psychiatric disorders, autoimmune disease, pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three hundred and eighty-eight patients were included in the study. One hundred and sixty-five were HCV genotype 1 subtype 1a (42.5%) while two hundred twenty-three were of subtype 1b (57.5%).
Sampling Method: Probability Sample
Enrollment: 388 (Actual)
Dates: Start 2007-02; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The primary end point was sustained undetectable serum HCVRNA 24 weeks after treatment cessation (SVR). | 24 weeks after treatment cessation
  The primary end point was sustained undetectable serum HCVRNA 24 weeks after treatment cessation (Sustained virological response).

CONTACTS AND LOCATIONS:
Overall Officials: Adriano M Pellicelli, MD, Study Director — AO Scamilloforlanini Rome Italy
Locations (1):
- AO San Camillo Forlanini, Rome, Italy, Italy

REFERENCES:
- [Derived] Pellicelli AM, Romano M, Stroffolini T, Mazzoni E, Mecenate F, Monarca R, Picardi A, Bonaventura ME, Mastropietro C, Vignally P, Andreoli A, Marignani M, D'Ambrosio C, Miglioresi L, Nosotti L, Mitidieri O, Gentilucci UV, Puoti C, Barbaro G, Barlattani A, Furlan C, Barbarini G; CLEO Group. HCV genotype 1a shows a better virological response to antiviral therapy than HCV genotype 1b. BMC Gastroenterol. 2012 Nov 16;12:162. doi: 10.1186/1471-230X-12-162. PMID 23157720
- See also: web site of AO SCamillo Forlanini Hospital — http://www.scamilloforlanini.rm.it